CLINICAL TRIAL: NCT05700136
Title: Prenatal and Postnatal Factors Associated With Infant Circadian Rhythm, Growth, and Temperament
Brief Title: Factors Associated With Infant Circadian Rhythm, Growth, and Temperament
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UCSI University (Other)
Responsible Party: Principal Investigator, Satvinder Kaur, Dr, UCSI University
Other Study IDs: RSCH ID-21-01830-S1K
Record Dates: First submitted 2023-01-05; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Circadian Rhythm Sleep Disorder, Jet Lag Type
Keywords: Circadian rhythm; Chrononutrition; Pregnancy; Infant; Eating misalignment; Light exposure
MeSH Terms: conditions — Jet Lag Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples Without DNA — Saliva samples were collected at third trimester and three months after birth for both mother and infant. Samples were analyzed to determine cortisol rhythm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MOMENT cohort: The cohort will be recruited at third trimester of pregnancy and required to fill up questionnaires and complete saliva collection. We will then follow up with the cohort at 3 months after birth to collect follow up data of the mother and infant. Lastly, we will collect growth outcomes of the infant at 6 months.
  Interventions: Behavioral: MOMENT

INTERVENTIONS:
Behavioral: MOMENT — Prenatal and postnatal factors including maternal, environment, and infant circadian rhythm were studied to determine its effect on infant growth and temperament.

SUMMARY:
The goal of this observational study is to learn about the role of modifiable factors affecting infant circadian rhythm so that recommendations can be made for better health outcomes for the mother and infant. The main questions it aims to answer are:

1. What is the association of prenatal and postnatal maternal circadian clock with infant's circadian clock at 3 months?
2. What is the association of birth outcomes, maternal factors, and environmental factors with infant circadian clock at 3 months?
3. What is the role of infant circadian clock on infant growth and temperament at 6 months of age?

Participants will complete a set of questionnaires and provide saliva samples during third trimester of pregnancy and at 3 months after birth of infant.

DETAILED DESCRIPTION:
Circadian rhythm is the body's internal clock that synchronizes the body's physiological functions according to the 24-hour sleep-wake cycle. An individual establishes a circadian rhythm 3 months after birth, which is a progressive phase that involves regulating hormones such as cortisol and melatonin. According to previous studies, the synchronization of circadian rhythm between mother-infant pairs have been found to be beneficial in the growth and development of the child by regulating a 24-hour sleep-wake cycle. However, circadian disruption may cause excessive maternal cortisol which can be transferred to the fetus through the placenta during pregnancy and cause growth retardation. Growth faltering during infancy is associated with increased risks of morbidity from infections and chronic diseases in later life. Therefore, it is important to study the relationship between maternal circadian rhythm with synchronization of infant circadian rhythm as it may be one of the potential factors which affects the growth and development of the child.

On the other hand, infant temperament is affected by the maternal and infant circadian rhythm and may also be a predictor to mood disorders such as depression and anxiety. A systematic review reported that high cortisol levels during third trimester of pregnancy is associated with higher emotional reactivity and more difficult temperament infants. Other than the biological factors determining infant temperament, maternal psychological wellbeing during and after pregnancy is also an important element. It has been found that elevated maternal stress was associated with negative infant temperament, resulting in decreased sleep quality of the infant. Negative infant temperament may be a predictor to disordered eating behaviors and growth development. As infant temperament is an important factor in determining growth and development, the risk factors to negative temperament should be studied.

This study aims to determine the role of prenatal and postnatal factors with the infant circadian rhythm and its relationship with infant growth and temperament at 6 months. This study also includes the validation of the Chrononutrition Profile Questionnaire (CPQ) among pregnant women. Through the validation of CPQ, future research about chrononutrition behaviors and eating misalignment can be conducted to replace food record. The design of this study is a prospective observational cohort study. Data will be collected during 3rd trimester of pregnancy, whereas follow-up data on birth outcomes will be collected at birth. At 3 months after birth, data on maternal and infant circadian rhythm will be assessed, then data on growth and development will be collected at 6 months after birth. Data collection is elicited through a properly designed and validated questionnaire namely Chrononutrition Profile Questionnaire (CPQ), Harvard Light Exposure Assessment (H-LEA), sun exposure habits, Morningness-Eveningness Questionnaire (MEQ), Positive and Negative Affect Schedule (PANAS), Pittsburgh Sleep Quality Index (PSQI), and Edinburgh Postnatal Depression Scale (EDPS). Meanwhile, anthropometric data such as gestational weight gain and birth outcomes are gathered from clinic record. In addition, data on infant sleep, feeding, behavior, and light exposure will be collected using Brief Infant Sleep Questionnaire (BISQ), infant feeding log, Baby Eating Behavior Questionnaire (BEBQ), Infant Behavior Questionnaire- Revised (IBQ-R), and infant light exposure log sheet. Cortisol levels will be determined using salivary cortisol method where maternal and infant saliva samples are collected at 3 time points: upon awakening, noon (10:00 to 12:00), and evening (19:30 to 21:00). Understanding the potential factors affecting infant circadian rhythm offers new insights in understanding modern lifestyle factors and its association with fetal programming, infant growth, and development.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women with no comorbidities before or during pregnancy
* Malaysian aged 18-39 years old
* Literate in English and Malay language
* Single pregnancy

Exclusion Criteria:

* Physically disabled
* Smoke cigarette and drinks alcohol during pregnancy
* On steroid medication
* Infants with any deformities or congenital diagnosis.

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is done among pregnant women only. Hence, only females were recruited in this study.
Study Population: The study population is pregnant women in third trimester from Kuala Lumpur, Malaysia. Pregnancy is a crucial timing where the nutrient intake of the mother contributes to the development of the child. Circadian rhythm during pregnancy may experience a change in phase as the cortisol release increases throughout pregnancy. While Malaysia faces the double burden of stunting and overweight among children, modernization has also caused various health consequences through circadian rhythm disruption, mainly by exposure to light at night and limited natural light exposure. Hence, pregnant women in Malaysia urban areas were studied.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Infant growth in height | Birth to 6 months
  Infant growth is determined by measuring the height (in centimeters) and height for age
Infant growth in weight | Birth to 6 months
  Infant growth is determined by measuring the weight (in kiligrams) and weight for age
Infant growth in head circumference | Birth to 6 months
  Infant growth is determined by measuring the head circumference (in centimeters)
Infant temperament | 6 months after birth
  Infant temperament is determined by completing the Infant Behavior Questionnaire- Revised version (IBQ-R)

SECONDARY OUTCOMES:
Infant circadian rhythm | 3 months after birth
  Infant circadian rhythm is determined by charting the cortisol rhythms that were tested using saliva samples

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Lian Aun In, Study Director — UCSI University
Locations (10):
- Malaysia (10):
  - Klinik Kesihatan Segambut, Kuala Lumpur
  - Klinik Kesihatan Metro Prima, Kuala Lumpur
  - Klinik Kesihatan Cheras Makmur, Kuala Lumpur
  - Klinik Kesihatan Kuchai Ent Park, Kuala Lumpur
  - Klinik Kesihatan Salak Selatan, Kuala Lumpur
  - Klinik Kesihatan Pantai Indah, Kuala Lumpur
  - Klinik Kesihatan Putrajaya Presint 11, Putrajaya
  - Klinik Kesihatan Putrajaya Presint 14, Putrajaya
  - Klinik Kesihatan Putrajaya Presint 18, Putrajaya
  - Klinik Kesihatan Putrajaya Presint 9, Putrajaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kok EY, Kaur S, Mohd Shukri NH, Abdul Razak N, Takahashi M. Development, validation, and reliability of the Chrononutrition Profile Questionnaire-Pregnancy (CPQ-P). BMC Pregnancy Childbirth. 2024 Mar 23;24(1):217. doi: 10.1186/s12884-024-06403-4. PMID 38521925